CLINICAL TRIAL: NCT05497310
Title: Effectiveness and Safety of Therapy Based on Attenuated Arsenic Trioxide Plus Low Doses of All-trans Retinoic Acid as Remission Induction Therapy in Patients With Acute Promyelocytic Leukemia Phase 1/2 Clinical Trial
Brief Title: Effectiveness and Safety of Therapy Based on Attenuated ATO Plus Low-Dose ATRA in Patients With APL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Head of Hematology Service, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE22-00019
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Promyelocytic Leukemia
Keywords: all-trans retinoic acid; arsenic trioxide; frontline therapy; induction chemotherapy
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide; Tretinoin

STUDY DESIGN:
Intervention Model Description: A consecutive sample of 15 patients with newly diagnosed or relapsed APL who have not been previously treated with ATO will be prospectively included in this study.
Masking Description: This is an Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction with attenuated ATO plus low-dose ATRA (Experimental): Remission induction therapy will be administrated as ATRA 25/mg/m2/day for 28 continuous days without interruption if APL is suspected. ATO 0.3mg/kg/day for days 1-5 (5 doses) and then 0.25 mg/kg/day every other day twice a week for the next 3 weeks (6 doses).
  Interventions: Drug: Arsenic trioxide; Drug: all-trans retinoic acid

INTERVENTIONS:
Drug: Arsenic trioxide — Patients will receive ATO 0.3mg/kg/day for days 1-5 (5 doses) and then 0.25 mg/kg/day every other day twice a week for the next 3 weeks (6 doses).
  Other Names: Trisenox
Drug: all-trans retinoic acid — Patients will receive ATRA 25/mg/m2/day for 28 continuous days without interruption.
  Other Names: Vesanoid

SUMMARY:
ATRA is the standard of care for all patients with APL. The use of lower doses of ATRA has been shown since the 1990s to achieve therapeutic efficacy with doses of 25mg/m2/day. ATO demonstrated considerable effectiveness in this disease. More recently, an attenuated regimen has been proven to be effective. In this study we intent to demonstrate the effectiveness of combined therapy of low-dose ATRA plus attenuated dose ATO.

DETAILED DESCRIPTION:
The use of lower doses of ATRA has been shown since the 1990s to achieve therapeutic plasma concentrations sufficient to achieve therapeutic efficacy with doses of 25mg/m2/day. ATO alone demonstrated considerable effectiveness in this disease. More recently, an attenuated regimen has been proven to be effective in inducing similar remission rates and achieving prolonged survival, also demonstrating a reduction in associated toxicities, mainly hepatic and cardiac when using this new scheme.

The investigators will conduct a phase 1/2, non-randomized, single center, non-comparative clinical trial to demonstrate the effectiveness of combined therapy of low-dose ATRA plus attenuated dose ATO which is accessible to a population with limited resources while maintaining acceptable efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Both genders
* new diagnosis of APL
* Diagnosis of relapsed APL who have not been previously treated with ATO
* Morphological diagnosis of APL confirmed by PCR or FISH

Exclusion Criteria:

* Poor functional status (ECOG>2)
* Organic dysfunction (Marshall score ≥2)
* Pregnancy
* Heart failure (NYHA III or IV)
* Renal failure (GFR <30 ml/min/1.72m2)
* History of ventricular arrhythmias or uncontrolled arrhythmias
* Acute myocardial infarction, unstable angina, or stable angina in the last six months
* Uncontrolled active infection
* Liver disease (Child-Pugh C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days
  Safety will be defined by the number of patients deceased after 1 induction cycle of 28 days

SECONDARY OUTCOMES:
Overall response | 28 days
  Overall response rate was definide as partial response plus complete response after 1
Progression-free survival | 6 months
  Time from achievement of complete hematologic remission to relapse
Event-free survival | 6 months
  Time from registration to induction failure, relapse, or death.
Rate of treatment discontinuation due to toxicity. | 28 days
  Rate of treatment discontinuation due to toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopsital Universitario Dr. Jose E. Gonzalez, Centro Universitario contra el Cancer, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang ME, Ye YC, Chen SR, Chai JR, Lu JX, Zhoa L, Gu LJ, Wang ZY. Use of all-trans retinoic acid in the treatment of acute promyelocytic leukemia. Blood. 1988 Aug;72(2):567-72. PMID 3165295
- [Background] Chen GQ, Zhu J, Shi XG, Ni JH, Zhong HJ, Si GY, Jin XL, Tang W, Li XS, Xong SM, Shen ZX, Sun GL, Ma J, Zhang P, Zhang TD, Gazin C, Naoe T, Chen SJ, Wang ZY, Chen Z. In vitro studies on cellular and molecular mechanisms of arsenic trioxide (As2O3) in the treatment of acute promyelocytic leukemia: As2O3 induces NB4 cell apoptosis with downregulation of Bcl-2 expression and modulation of PML-RAR alpha/PML proteins. Blood. 1996 Aug 1;88(3):1052-61. PMID 8704214
- [Background] Castaigne S, Lefebvre P, Chomienne C, Suc E, Rigal-Huguet F, Gardin C, Delmer A, Archimbaud E, Tilly H, Janvier M, et al. Effectiveness and pharmacokinetics of low-dose all-trans retinoic acid (25 mg/m2) in acute promyelocytic leukemia. Blood. 1993 Dec 15;82(12):3560-3. PMID 8260694
- [Background] Chen GQ, Shen ZX, Wu F, Han JY, Miao JM, Zhong HJ, Li XS, Zhao JQ, Zhu J, Fang ZW, Chen SJ, Chen Z, Wang ZY. Pharmacokinetics and efficacy of low-dose all-trans retinoic acid in the treatment of acute promyelocytic leukemia. Leukemia. 1996 May;10(5):825-8. PMID 8656678
- [Background] Jaime-Perez JC, Gonzalez-Leal XJ, Pinzon-Uresti MA, Gomez-De Leon A, Cantu-Rodriguez OG, Gutierrez-Aguirre H, Gomez-Almaguer D. Is There Still a Role for Low-Dose All-Transretinoic Acid in the Treatment of Acute Promyelocytic Leukemia in the Arsenic Trioxide Era? Clin Lymphoma Myeloma Leuk. 2015 Dec;15(12):816-9. doi: 10.1016/j.clml.2015.09.002. Epub 2015 Sep 25. PMID 26500134
- [Background] Burnett AK, Russell NH, Hills RK, Bowen D, Kell J, Knapper S, Morgan YG, Lok J, Grech A, Jones G, Khwaja A, Friis L, McMullin MF, Hunter A, Clark RE, Grimwade D; UK National Cancer Research Institute Acute Myeloid Leukaemia Working Group. Arsenic trioxide and all-trans retinoic acid treatment for acute promyelocytic leukaemia in all risk groups (AML17): results of a randomised, controlled, phase 3 trial. Lancet Oncol. 2015 Oct;16(13):1295-305. doi: 10.1016/S1470-2045(15)00193-X. Epub 2015 Sep 14. PMID 26384238